CLINICAL TRIAL: NCT04661098
Title: Formation of an Annular Hymen in Cases of Postpubertal Imperforate Hymen Using a Laparoscopic Trocar (Darwish Hymenotomy Technique)
Brief Title: Darwish Hymenotomy Technique in Cases of Postpubertal Imperforate Hymen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Atef Darwish (Other)
Responsible Party: Sponsor-Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Organization: Woman's Health University Hospital, Egypt (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Darwish hymenotomy technique
Record Dates: First submitted 2020-05-19; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Imperforate Hymen
Keywords: imperforate; hymenotomy; annular; laparoscopic; trocar; postpubertal; hymen
MeSH Terms: conditions — Hymen, Imperforate

STUDY DESIGN:
Intervention Model Description: Formation of an annular hymen in cases of postpubertal imperforate hymen using a laparoscopic trocar (Darwish hymenotomy technique)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Postpubertal patients with imperforate hymen (Experimental): Formation of an annular hymen in cases of postpubertal imperforate hymen using a laparoscopic trocar (Darwish hymenotomy technique)
  Interventions: Procedure: (Darwish hymenotomy technique)

INTERVENTIONS:
Procedure: (Darwish hymenotomy technique) — Formation of an annular hymen in cases of postpubertal imperforate hymen using a laparoscopic trocar (Darwish hymenotomy technique)

SUMMARY:
This study aims to test the use of a 10 mm laparoscopy trocar tip for formation of a new vaginal orifice with preservation of an annular hymen (Darwish hymenotomy technique) in cases of post pubertal imperforate hymen (IH). A prospective interventional case series done at a minimally invasive surgery unit of a tertiary university hospital between July 2013 and October 2019 comprising patients with primary amenorrhea and hematocolpus. Circular hymenotomy using a 10 mm laparoscopy trocar tip and sleeve done under general anesthesia was done in 36 cases. Documented vaginal patency with formation of an annular hymen in all cases was reported on follow-up visits without reported intraoperative complications. Patient and family satisfaction with excellent sensation of preserved hymen was also documented. Using a 10 mm laparoscopy trocar tip for formation of a new vaginal opening with preservation of annular hymen (Darwish technique) in cases of postpubertal IH is a simple, effective and safe procedure suitable for Islamic and conservative societies with excellent impact on the psychological and emotional status of the patient and her family.

DETAILED DESCRIPTION:
This study is a prospective interventional case series conducted at the Minimally Invasive Surgery Unit of the Woman's Health University Hospital, Assiut, Egypt, between July 2013 and October 2019. It was approved in May 2013 by the local ethical committee of the faculty of Medicine, Assiut University. After detailed explanation of the study, all cases or parents signed an informed consent to participate in this study. It comprised 43 cases with primary amenorrhea and hematocolpus. Patients' complaints included a gradually progressive central abdominal mass, pelvic pain getting worse over time disturbing her studies, urinary retention, dysuria, constipation and dyschezia separately or collectively depending on the chronicity of retained menstruation. Clinical examination started by downward labial traction to separate the labia majora and minora sufficiently to visualize the distal introitus. Girls with only IH as diagnosed after puberty (postpubertal) without any suspicion of associated congenital anomaly were included in this study. Low transverse vaginal septum was diagnosed in 4 cases that were excluded from this study. Differentiation between IH and transverse vaginal septum relied mainly on clinical examination in the lithotomy position with insertion of a uterine sound into the dimple. If the sound fails to go up, it is a case of IH. If it goes up this means a low transverse vaginal septum that requires an advancement operation with fixation of the edges of the septum to the introitus. In such cases, hymentomy will fail with reformation of the septum as it is thick in contrast to the thin hymen. During examination, distal vaginal atresia was excluded by the absence of hymnal distension on Valsalva and absence of its bluish discoloration in addition to far existence of the hematocolpos away from the vulva. It was reported in two cases that were also excluded from the study. If the abdominal mass was noticed to be deviated to one side, a possibility of type I obstructed hemi-vagina and ipsilateral renal agenesis (OHVIRA) raised and a confirmatory MRI was requested. Only one case with OHVIRA type I (Blind hemi-vaginal septum without an opening) was detected and excluded from the study. This case presented with primary amenorrhea due to a rudimentary contralateral horn. Clinical examination of 36 cases with IH was relatively easy as the patient presented with a vaginal bulge of thin hymenal tissue with a dark or bluish hue caused by the hematocolpos behind it. If the physical examination revealed a bulging hymen and ultrasonography confirmed the diagnosis of hematocolpos, further imaging was not required. In selected cases with ambiguous diagnosis, MRI was requested to assess the vaginal and the perineum in a meticulous way. For surgical safety, prepubertal girls with IH were excluded.

The procedure stars by putting the patient in the lithotomy position in the OR. After induction of general anesthesia, sterilization and toweling of the perineum was done. Insertion of an indwelling urethral catheter and PR to exclude other anomalies or abnormalities were done. The tip of a 10 mm laparoscopy trocar with a sharp triangular point (Karl Storz, Tuttlingen, Germany) was inserted in the center of the most bulging point of the IH. Once the edge of the sleeve followed the tip of the trocar tip into the hymen, no further advancement of the trocar tip was made to avoid unintentional injuries by the trocar itself. After its withdrawal, the sleeve was left insitu for drainage of the retained blood. Suprapubic pressure was not done to avoid ascending infection by the negative pressure. After complete stoppage of flow of the retained menstruation the sleeve was removed. Usually no further intervention was needed. If oozing points were seen, a gentle bipolar coagulation was used. The remaining hymenal ring was evaluated and documented in the patient's file whether intact circular or not. All technical steps are shown in figure 1. After recovery, the patient was kept for few hours in the postoperative ward then discharged. She was advised to come for follow-up after the coming menstruation or after 40 days if no menses occur. She was examined to ensure patency of the vagina, the integrity of the hymen and sonographically to ensure absence of retained menstruation and to assess both kidneys. Subsequent follow-up visits were optional whenever they notice any change in the menstrual flow. Otherwise telephone calls were kept with them thereafter. Outcomes included hymenal ring integrity on naked eye examination, patient satisfaction, relief of symptoms, and a feeling of well-being. Due to rarity of cases, the same patient was used to compare preoperative and postoperative results.

ELIGIBILITY:
Inclusion Criteria: postpubertal imperforate hymen

-

Exclusion Criteria:

* Prepubertal imperforate hymen

Ages: 12 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Hymenal patency | 1 month
  examination postoperatively to see opened hymen.
Integrity | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Atef Darwish, Principal Investigator — Woman's Health University Hospital

IPD SHARING:
Plan to Share IPD: No